CLINICAL TRIAL: NCT00324454
Title: A Pilot Trial of Levetiracetam for Cramps, Spasticity and Neuroprotection in Motor Neuron Disease
Brief Title: Levetiracetam for Cramps, Spasticity and Neuroprotection in Motor Neuron Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00005846; 8380-06-3R0 (Other: DUMC)
Record Dates: First submitted 2006-05-09; First posted 2006-05-11 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2009-01

CONDITIONS: Motor Neuron Disease; Amyotrophic Lateral Sclerosis; Primary Lateral Sclerosis; Progressive Muscular Atrophy
Keywords: motor neuron disease; amyotrophic lateral sclerosis primary lateral; sclerosis; progressive muscular atrophy; cramps; spasticity
MeSH Terms: conditions — Motor Neuron Disease; Amyotrophic Lateral Sclerosis; Muscular Atrophy, Spinal; Sclerosis; Muscle Cramp; Muscle Spasticity | interventions — Levetiracetam; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Levetiracetam — Levetiracetam 1500 mg BID
  Other Names: Keppra 1500 mg BID

SUMMARY:
Levetiracetam (Keppra) is used to treat partial onset seizures. Its biological effects suggest it might also be useful in treating 3 aspects of human motor neuron diseases (MNDs) for which no effective therapy exists: cramps, spasticity, and disease progression.

DETAILED DESCRIPTION:
Cramps in MNDs are believed to occur as a result of high-frequency burst firing of alpha motor neurons. Levetiracetam inhibits burst firing in epileptic rat hippocampus. Levetiracetam has never been tested against cramps in humans; however, it has helped another condition believed to result from burst firing of a motor nerve: hemi-facial spasm.

The mechanisms underlying spasticity in MNDs likely involve imbalance between excitatory and inhibitory influences on the alpha motor neurons. Levetiracetam may modulate these influences in a number of ways, including reducing the effects of zinc and beta-carbolines in GABA and glycine receptors. Levetiracetam reduces phasic (but not tonic) spasticity in patients with multiple-sclerosis.

Levetiracetam may have neuroprotective properties. In a model of cerebral ischemia induced by occlusion of the rat internal carotid artery, pre-treatment with levetiracetam reduced infarct size in a dose-dependent manner. In rats injected with kainic acid to induce calcium overload, oxidative stress and neurotoxicity, pretreatment with levetiracetam offset kainic acid's effects. The mechanisms for these effects may relate to levetiracetam's ability to influence calcium currents, or its ability to increase the release of growth factors from astrocytes, mechanisms that would be relevant in MNDs. Levetiracetam's ability to inhibit histone deacetylase may also help slow MNDs progression.

OBJECTIVES: 1. Assess the safety and tolerability of levetiracetam over 9 months in patients with MNDs. 2. Determine whether treatment with levetiracetam is associated with a reduction in cramps, spasticity or motor neuron disease progression.

METHODS:Open-label, Phase 2 trial of 20 adult patients with MNDs (ALS, PLS or PMA) at Duke University ALS Clinic. Eligible patients have cramps with average severity 50/100 points, are able to provide informed consent, have normal renal functions and are on a stable riluzole dose. Exclusions include pregnancy, unstable mental illness, dementia, drug abuse or non-compliance. The first 3 months of the study are a baseline period. Over the remaining 9 months, patients take levetiracetam at increasing doses up to 3000mg per day. Outcome measures include adverse events, tolerability,cramp-pain-severity score, cramp-frequency score, modified Ashworth Spasticity Score, Penn Spasm Score, FVC, ALSFRS-R and MMT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with MNDs (ALS, PLS or PMA)who have cramps with average severity 50/100 points, are able to provide informed consent, have normal renal function and are on a stable riluzole dose.

Exclusion Criteria:

* Pregnancy; unstable medical illness, dementia; drug abuse or non-compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-05; Primary Completion 2007-12 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability at 9 months of treatment. | 9 months

SECONDARY OUTCOMES:
Cramps scores, spasticity scores, FVC, ALSFRS, MMT | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Bedlack, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University ALS Clinic - 932 Morreene Road, Durham, North Carolina, United States